CLINICAL TRIAL: NCT05366322
Title: Real-world Comparative Effectiveness of the mRNA-1273 Vaccine vs. BNT162b2 Vaccine Among Immunocompromised Adults in the United States
Brief Title: A Study to Compare mRNA-1273 Versus BNT162b2 COVID-19 Vaccines Among Immunocompromised Adults
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P913
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort A: mRNA-1273 COVID Vaccine: Participants who have received 2 doses of the mRNA-1273 vaccine at least 14 days apart.
- Cohort B: BNT1262b2 COVID Vaccine: Participants who have received 2 doses of the BNT1262b2 vaccine at least 14 days apart.

SUMMARY:
The goal of this study is to compare real-world effectiveness of the mRNA-1273 vaccine versus the BNT162b2 vaccine on medically attended COVID-19 and COVID-19 hospitalizations among fully vaccinated immunocompromise participants.

DETAILED DESCRIPTION:
This observational retrospective comparative effectiveness cohort study will use the HealthVerity aggregated medical and pharmacy claims database. HealthVerity data elements include provider-submitted claims, adjudicated insurance claims, and pharmacy billing manager claims submissions. Hospitalizations are included in the data at a summary level.

ELIGIBILITY:
Inclusion Criteria:

* Fully vaccinated with a currently US authorized COVID-19 vaccine:
* 2 doses of mRNA-1273 (minimum 14 days between doses)
* 2 doses of BNT1262b2 (minimum 14 days between doses)
* Continuous enrollment in medical & pharmacy plan for at least 365 days prior to index/Cohort entry date (CED)
* Identified as immunocompromised via at least 1 of the following criteria at index/CED
* Evidence of blood or stem cell transplant in 2 years prior to index/CED
* Any history of organ transplant and taking immunosuppressive therapy within the 60 days prior to index/CED
* Evidence of active cancer treatment in the 180 days prior to index/CED with an active cancer diagnosis in the 365 days prior to treatment
* Any prior history of a primary immunodeficiency disorder (for example, for conditions such as DiGeorge syndrome and Wiskott-Aldrich syndrome)
* Any history of an HIV diagnosis code prior to index/CED
* A fill for an immunosuppressive therapy in the 60 days prior to index/CED

Exclusion Criteria:

* Prior COVID-19 infection (any history prior to index/CED through day 13 post-completion of vaccine regimen) identified via the following diagnosis codes on an inpatient or outpatient claim:
* U07.1: "COVID-19, virus identified"
* J12.82: "Pneumonia due to COVID-19"
* Z86.16: "Personal history of COVID-19"
* The following diagnosis codes were utilized early in the pandemic. Exclusion will be applied March 1, 2020 through day 13 post-completion of vaccine regimen:
* J12.89: "Other viral pneumonia"
* J20.8: "Acute bronchitis due to other specified organisms"
* J40: "Bronchitis, not specified as acute or chronic"
* J22: "Unspecified acute lower respiratory infection"
* J98.8: "Other specified respiratory disorders"
* J80: "Acute respiratory distress syndrome"
* Prior receipt of a heterologous COVID-19 vaccine (relative to the COVID-19 vaccine identified at index/CED) in the 365 days prior to index/CED through 13 days post-completion of vaccine regimen
* Receipt of an additional dose of homologous COVID-19 vaccine between index/CED and 13 days post-completion of vaccine regimen
* Missing or unknown gender on index/CED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from HealthVerity's aggregated medical and pharmacy claims database that represents healthcare utilization for participants between 01 December 2018 and 10 January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 124879 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Medically Attended Breakthrough COVID-19 Diagnosis | Index date (14-days post-receipt of 2nd dose of mRNA-1273 to BNT162b2) up to end of available data (12 October 2021 [up to 9 months])
  Medically attended breakthrough COVID-19 diagnosis defined as a claim for COVID-19 in any setting (inpatient, outpatient, emergency room, urgent care, etc.).

SECONDARY OUTCOMES:
Number of Participants with Breakthrough Hospitalization for COVID-19 | Index date (14-days post-receipt of 2nd dose of mRNA-1273 to BNT162b2) up to end of available data (12 October 2021 [up to 9 months])
  Breakthrough hospitalization for COVID-19 defined as a hospital stay for COVID-19 listed as the primary diagnosis or within 21 days prior to hospital admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Aetion Inc., New York, New York, United States

REFERENCES:
- [Derived] Mues KE, Kirk B, Patel DA, Gelman A, Chavers LS, Talarico CA, Esposito DB, Martin D, Mansi J, Chen X, Gatto NM, Van de Velde N. Real-world comparative effectiveness of mRNA-1273 and BNT162b2 vaccines among immunocompromised adults identified in administrative claims data in the United States. Vaccine. 2022 Nov 8;40(47):6730-6739. doi: 10.1016/j.vaccine.2022.09.025. Epub 2022 Sep 24. PMID 36163093